CLINICAL TRIAL: NCT00633529
Title: Open-Label Phase 1b Study of Erlotinib Plus Bevacizumab and IMO-2055 in Patients With Non-Small Cell Lung Cancer Who Have Progressed Following Initial Chemotherapy for Advanced or Metastatic Disease
Brief Title: Safety of Adding IMO-2055 to Erlotinib + Bevacizumab in 2nd Line Treatment for Patients With NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: EMR 200068-200
Record Dates: First submitted 2008-03-03; First posted 2008-03-12 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Phase 1b; Non-Small Cell Lung Cancer; Advanced or Metastatic Disease; Prior chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — IMO-2055

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Single arm: triple combination
  Interventions: Drug: IMO-2055

INTERVENTIONS:
Drug: IMO-2055 — 0.08, 0.16, or 0.32 mg/kg SC (subcutaneous) on days 1,8,and 15 of every 21 day cycle until evidence of progressive disease, unacceptable treatment-related toxicities, withdrawal of patient consent and/or Investigator decision to withdraw study therapy with documented reason, whichever occurs first.

SUMMARY:
To evaluate the safety of the proposed Phase II dosage of the investigational drug IMO 2055 when combined with erlotinib and bevacizumab in patients with previously treated advanced NSCLC.

DETAILED DESCRIPTION:
Phase 1b study of escalating doses of weekly subcutaneous IMO-2055 combined with fixed standard dose regimens of oral erlotinib (daily) and IV bevacizumab (every 3 weeks) in patients with previously treated advanced NSCLC.

ELIGIBILITY:
Inclusion:

Patients must satisfy all the following inclusion criteria in order to be eligible for the study:

1. Signed written informed consent
2. AJCC stage 3 or 4 histologically proven NSCLC not amenable to curative therapy and for whom erlotinib and bevacizumab therapy would be appropriate
3. Radiological assessment within 21 days prior to inclusion, if measurable disease is present
4. Age ≥ 18 years
5. ECOG performance status 0 or 1
6. Patient has received at least one standard platinum-containing chemotherapy regimen appropriate for his/her lung cancer, in the opinion of the investigator, prior to enrollment.

Exclusion:

Patients with any of the following will be excluded from participation in the study:

Disease

1. Squamous cell carcinoma, except for patients with no intrathoracic disease or small peripheral lesions only.
2. Known central nervous system (CNS) metastases (Note: patients with brain metastases which have been controlled for ≥ 4 months without the use of steroid are eligible).

   Prior Treatments
3. Less than 4 weeks between registration and the last receipt of chemotherapy, biotherapy, radiotherapy or major surgery
4. Concurrent or planned hormonal agents such as replacement therapy, oral contraceptives, or anti-cancer therapy, e.g. Megace. (A prior history of such therapy is not exclusionary.)
5. Administration of any investigational agent (therapeutic or diagnostic), including any investigational compound for the treatment of NSCLC, within 4 weeks prior to first study dosing Other Concomitant Medications
6. High dose oral or intravenous corticosteroids. (Note: topical, inhaled and intra-articular corticosteroids are allowed. Prophylactic antihistamines are allowed before administration of bevacizumab
7. Use of any medication which is a strong inhibitor or inducer of cytochrome P450 isoform CYP3A4 (see Appendix 5)
8. Therapeutic dosing with warfarin >1 mg/day
9. Chronic daily use of aspirin (> 325 mg/day) or other full-dose NSAIDs with anti-platelet activity
10. Inability to take oral medication or requirement for IV alimentation or total parenteral nutrition with lipids, or prior surgical procedures affecting absorption Laboratory
11. The following laboratory results, within 10 days of first study drug administration:

    * Hemoglobin ≤ 9.0 g/dL Absolute neutrophil count ≤ 1.5 x 109/L Platelet count ≤ 100 x 109/L
    * International Normalized Ratio (INR) > 1.3 (only if the subject is on warfarin [< 1 mg per day]) during 28 days prior to enrollment.
    * aPTT > Upper Limit of Normal (ULN) during 28 days prior to enrollment.
    * Serum creatinine ≥ 1.5 x ULN and creatinine clearance (by Cockcroft-Gault formula) <60 mL/min
    * Serum bilirubin ≥ 1.5 x ULN
    * Proteinuria: UPC ≥ 1.0 or ≥ 2+ proteinuria by urine dipstick, unless a 24-hour urine demonstrates <1.0 g/24 hours
    * ALT or AST ≥ 2.5 x ULN (≥ 5 x ULN if liver metastases)
    * Alkaline phosphatase ≥ 2.5 x ULN
    * Albumin ≤ 2.5 g/L
    * Women of child bearing potential: positive pregnancy test (serum). Other Conditions or Procedures
12. Any clinically significant adverse events from any prior chemotherapy, surgery or radiotherapy which has not yet resolved to CTCAE v3.0 grade ≤ 1
13. Known hypersensitivity to any oligodeoxynucleotide (ODN), EGFR-inhibitor or bevacizumab
14. Serious, non-healing wound, ulcer or bone fracture
15. Patients with a history or current neoplasm other than the entry diagnosis, except for curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix and except for other cancers treated for cure and with a disease-free survival greater than 5 years.
16. Pregnant or breast-feeding women
17. Men or women of childbearing potential who refuse or who are unable to use an acceptable means of contraception
18. History of clinically significant hemoptysis within 3 months prior to registration unless definitively treated with surgery or radiation
19. Any medical conditions that would impose excessive risk to the patient, such as uncontrolled hypertension (systolic >150 mmHg or diastolic >100 mmHg per JNC 7 guidelines, congestive heart failure NYHA Class 2-4, uncontrolled or unstable angina, myocardial infarction within the previous 6 months, ventricular arrhythmia, infection requiring parental or oral anti-infective treatment, any altered mental status or any psychiatric condition that would interfere with understanding the informed consent, uncontrolled seizures, chronic hepatitis or cirrhosis, known human immunodeficiency virus (HIV) infection, known hepatitis B surface antigen (HBsAg) positive or uncontrolled diabetes. (Note: testing for HIV infection of HBsAg is not part of the screening assessments performed by the central laboratory).
20. Pre-existing autoimmune or antibody-mediated diseases, including, but not limited to, the following: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome and autoimmune thrombocytopenia
21. Evidence of bleeding diathesis or coagulopathy or other serious or acute internal bleeding within 6 months prior to registration
22. CNS bleeding; history or clinical evidence of CNS stroke (hemorrhagic or thrombotic) within the last 6 months
23. History of allogeneic organ transplant
24. Brain biopsy within 12 weeks of first study dosing
25. Minor surgical procedure, central venous catheter placement, fine needle aspirations or core biopsy within 7 days prior to first study dosing
26. Anticipation of need for a major surgical procedure during the course of the study Other
27. Unwilling or unable to comply with the protocol for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To determine the recommended dosage of IMO-2055 when combined with erlotinib and bevacizumab in patients with AJCC stage 3 or 4 histologically proven non-small cell lung cancer (NSCLC). | Assessed on a weekly basis at patient visits.

SECONDARY OUTCOMES:
To evaluate the safety of weekly IMO-2055 combined with erlotinib plus bevacizumab using NCI CTCAE version 3. | Assessed on a weekly basis at patient visits.
To investigate potential drug-drug interactions via a PK study, specifically the effect of IMO-2055 on the PK of bevacizumab and the PK of erlotinib and also the effect of bevacizumab and erlotinib on the PK of IMO-2055. | Assessed on a weekly basis at patient visits.
To investigate potential signs of efficacy using RECIST response rate in measurable patients and PFS in all patients. | Assessed every six weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Breitfeld, MD, Study Director — EMD Serono
Locations (9):
- United States (9):
  - Cancer Centers of Florida, Ocoee, Florida
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - New York Oncology Hematology P.C., Albany, New York
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Shore Cancer Lodge, Yakima, Washington

REFERENCES:
- [Result] Smith, D., P. Conkling, D. Richards, C. Alemany, T. Boyd, L. Garbo, D. Loesch, D. Wages, A. Bexon, J. Murphy. Phase 1 Study of the Toll-like Receptor (TLR9) Agonist, IMO-2055, Combined with Erlotinib and Bevacizumab in Patients with Advanced or Metastatic non-Small Cell Lung Cancer. ECCO-ESMO Annual Meeting, 2009. Abstract 9.148.